CLINICAL TRIAL: NCT00000192
Title: Neurobiology of Opioid Dependence: 1
Brief Title: Neurobiology of Opioid Dependence: 1 - 1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00191-1; K20DA000191 (NIH); K20-00191-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Opioid-Related Disorders
Keywords: opioid disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine

SUMMARY:
The purpose of this study is to evaluate the effects of lamotrigine on naloxone-precipitated opiate withdrawal.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1993-01; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Behavioral, subjective, measures of naloxone-precipitated opiate withdrawal
Phsyiological, neuroendocrine measures of naloxone-precipitated opiate withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Rosen, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States

REFERENCES:
- [Background] Rosen MI, Pearsall HR, Kosten TR. The effect of lamotrigine on naloxone-precipitated opiate withdrawal. Drug Alcohol Depend. 1998 Oct 1;52(2):173-6. doi: 10.1016/s0376-8716(98)00057-x. PMID 9800147